CLINICAL TRIAL: NCT01287637
Title: Early Closure of Temporary Ileostomy- a Randomized Clinical Trial
Brief Title: Early Closure of Temporary Ileostomy
Acronym: EASY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Anne Kjærgaard Danielsen, Research Nurse, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKD03
Record Dates: First submitted 2011-01-28; First posted 2011-02-01 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Temporary ileostomy; Ealy reversal; Morbidity; Mortality; Quality of life; Economic effect
MeSH Terms: conditions — Rectal Neoplasms | interventions — Postoperative Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early reversal group (Experimental): Early reversal of temporary ileostomy
  Interventions: Procedure: Early reversal of temporary ileostomy
- Control group (Active Comparator): Standard reversal of temporary ileostomy
  Interventions: Procedure: Standard reversal of temporary ileostomy

INTERVENTIONS:
Procedure: Early reversal of temporary ileostomy — Temporary ileostomy is reversed 8-13 days after the primary surgery
  Other Names: stoma reversal 8-13 days post surgery
  Arms: Early reversal group
Procedure: Standard reversal of temporary ileostomy — Patients in the control group will have the ileostomy reversed according to standard treatment, which is 12-26 weeks after primary operation
  Other Names: stoma reversal 12-26 weeks after stoma creation
  Arms: Control group

SUMMARY:
The study is being conducted as a prospective randomized controlled multicenter study of patients with a temporary ileostomy due to rectal cancer. The study will be conducted in hospitals in Denmark and Sweden under the framework of the Scandinavian Surgical Outcomes Group (www.ssorg.net).

The study investigates the effect of reversing a temporary ileostomy after 8-13 days instead of later reversal more than 12 weeks after surgery.

DETAILED DESCRIPTION:
After creation of the temporary ileostomy patients are included and are randomized to two groups. Patients in the intervention group will have the stoma closed 8-13 days after stoma creation and will be compared to patients in the control group where the stoma is closed after a minimum of 12 weeks (standard treatment in Denmark and Sweden).

Before randomization the eligible patients undergo a CT of the rectum to visualise the anastomosis and possible leakage. Furthermore, the local investigators may choose to supplement the CT with a rectoscopy.

The research group includes 89 patients over an expected period of 4 years. Both groups are examined for postoperative complications as well as stoma-related complications at discharge and 3, 6 and 12 months after stoma creation.

The research group also examines the impact on patients´ health-related quality of life at 3, 6 and 12 months after stoma creation.

Finally the socio-economic effect in both groups will be analyzed and compared 6 and 12 months after stoma creation.

An interim analysis is planned for safety as well as recalculation of statistical power.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a temporary ileostomy after low anterior resection because of rectal cancer
* Patients, who are physically and mentally fit to undergo surgery within 8-13 days

Exclusion Criteria:

* Patients whose stoma is not reversible
* Patients with diabetes
* Patients being treated with Steroids
* Patients with communicative problems
* Patients with expected compliance issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2011-02; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Postsurgical morbidity | 3 months after inclusion
  Patients are scored according to the Clavien-Dindo Classification of Surgical Complications.
Postsurgical morbidity | 6 months after inclusion
  Patients are scored according to the Clavien-Dindo Classification of Surgical Complications.
Postsurgical morbidity. | 12 months after inclusion-
  Patients are scored according to the Clavien-Dindo Classification of Surgical Complications.

SECONDARY OUTCOMES:
Quality of life | Quality of life is assessed at 3 months after inclusion
  Patients quality of life is assessed with three questionnaires that supplement each other: Short Form 36 (SF-36), Ostomy Adjustment Scale (OAS) and European Organization for the Treatment of Cancer CR30+CR29 (EORTC QLQ-CR30+CR29)
Quality of life | Quality of life is assessed at 6 months after inclusion
  Patients quality of life is assessed with three questionnaires that supplement each other: Short Form 36 (SF-36), Ostomy Adjustment Scale (OAS) and European Organization for the Treatment of Cancer CR30+CR29 (EORTC QLQ-CR30+CR29)
Quality of life | Quality of life is assessed at 12 months after inclusion
  Patients quality of life is assessed with three questionnaires that supplement each other: Short Form 36 (SF-36), Ostomy Adjustment Scale (OAS) and European Organization for the Treatment of Cancer CR30+CR29 (EORTC QLQ-CR30+CR29)
Socio-economic effect of early reversal of temporary ileostomy | The investigators assess and analyze the economic effect 6 months after inclusion
  The investigators register all admissions to hospital and out-patient clinics up to 12 months after the operation. Furthermore, the investigators apply patients´self-reported data on visits to general practitioner, primary care nurses and other health care workers in primary care.
Socio-economic effect of early reversal of temporary ileostomy | The investigators assess and analyze the economic effect 12 months after inclusion
  The investigators register all admissions to hospital and out-patient clinics up to 12 months after the operation. Furthermore, the investigators apply patients´self-reported data on visits to general practitioner, primary care nurses and other health care workers in primary care.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Rosenberg, Professor, Principal Investigator — Herlev Hospital, University of Copenhagen
Locations (1):
- Herlev Hospital, University of Copenhagen, Herlev, Denmark

REFERENCES:
- [Derived] Park J, Angenete E, Bock D, Correa-Marinez A, Danielsen AK, Gehrman J, Haglind E, Jansen JE, Skullman S, Wedin A, Rosenberg J. Cost analysis in a randomized trial of early closure of a temporary ileostomy after rectal resection for cancer (EASY trial). Surg Endosc. 2020 Jan;34(1):69-76. doi: 10.1007/s00464-019-06732-y. Epub 2019 Mar 25. PMID 30911920
- [Derived] Park J, Danielsen AK, Angenete E, Bock D, Marinez AC, Haglind E, Jansen JE, Skullman S, Wedin A, Rosenberg J. Quality of life in a randomized trial of early closure of temporary ileostomy after rectal resection for cancer (EASY trial). Br J Surg. 2018 Feb;105(3):244-251. doi: 10.1002/bjs.10680. Epub 2017 Nov 23. PMID 29168881
- [Derived] Danielsen AK, Park J, Jansen JE, Bock D, Skullman S, Wedin A, Marinez AC, Haglind E, Angenete E, Rosenberg J. Early Closure of a Temporary Ileostomy in Patients With Rectal Cancer: A Multicenter Randomized Controlled Trial. Ann Surg. 2017 Feb;265(2):284-290. doi: 10.1097/SLA.0000000000001829. PMID 27322187
- [Derived] Danielsen AK, Correa-Marinez A, Angenete E, Skullmann S, Haglind E, Rosenberg J; SSORG (Scandinavian Outcomes Research Group). Early closure of temporary ileostomy--the EASY trial: protocol for a randomised controlled trial. BMJ Open. 2011 Jul 29;1(1):e000162. doi: 10.1136/bmjopen-2011-000162. PMID 22021780